CLINICAL TRIAL: NCT00598130
Title: A Prospective, Randomized, Single-Blind, Standard Care Controlled, Multi-Center, Phase II Study Evaluating the Safety and Hemostatic Efficacy of Fibrin Fleece in Partial Nephrectomy
Brief Title: Safety and Hemostatic Efficacy of Fibrin Fleece in Partial Nephrectomy
Acronym: Fleece
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OMRIX Biopharmaceuticals (Industry)
Responsible Party: Eran Kurman - Clinical Affaires Manager, Omrix Biopharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FL-PN-002-IS; MoH
Record Dates: First submitted 2007-12-23; First posted 2008-01-18 (Estimated); Last update posted 2009-11-06 (Estimated); Status verified 2009-11

CONDITIONS: Hemostatic Techniques; Nephrectomy
Keywords: Patients undergoing elective open partial nephrectomy surgery; Excision of a kidney
MeSH Terms: interventions — Collagen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Experimental): patients who will be treated in accordance with standard of care
  Interventions: Biological: Fleece
- II (Active Comparator): patients for which the Fibrin Fleece will be applied directly on the active bleeding site.
  Interventions: Biological: Fleece

INTERVENTIONS:
Biological: Fleece — Fibrin Patch

SUMMARY:
This is a prospective, randomized, single blind, standard care- controlled study, which will include a total of 30 patients divided into two treatment arms: First are: patents who will be treated in accordance with standard of care. Second arm: patients for which the Fibrin Fleece will be applied directly on the active bleeding site.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective open partial nephrectomy
* Patients must be willing to participate in the study, and provide written informed consent

Exclusion Criteria:

* Patients with a tumor diameter greater than 4 cm
* Any additional surgical intervention other than partial nephrectomy
* Patients with only one functional kidney
* Patients with known intolerance to blood products or other components of the product

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-11 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Proportion of successes at 10 minutes following randomization | 10 minutes

SECONDARY OUTCOMES:
Proportion of successes at 5 minutes following randomization | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Dekel, MD, Principal Investigator — Rabin MC
Locations (4):
- Israel (4):
  - Bnei-Zion MC, Haifa
  - Meir MC, Kfar Saba
  - Rabin MC, Tel Aviv
  - Sheaba MC, Tel Aviv

REFERENCES:
- [Derived] Nativ O, Patel B, Shen J, Batiller J, Horn S, Hart JC. Safety and hemostatic efficacy of fibrin pad in partial nephrectomy: results of an open-label phase I and a randomized, standard-of-care-controlled phase I/II study. BMC Nephrol. 2012 Nov 8;13:147. doi: 10.1186/1471-2369-13-147. PMID 23137020